CLINICAL TRIAL: NCT00468975
Title: A Phase IIA Randomised, Double-blind, Double Dummy, Placebo and Active Controlled 5-Way Cross-over Trial to Examine the Bronchodilator Effects of PF-610,355 and to Test for Superiority Versus Placebo in Reversible Asthmatic Patients
Brief Title: A Blinded Study To Examine The Ability Of PF-610,355 To Open The Airways In Asthmatic Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A7881004
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate

INTERVENTIONS:
Drug: PF-610,355
Drug: Salmeterol

SUMMARY:
A study to determine the ability of different doses of PF-610,355 to open the airways in asthmatic patients by comparison with placebo and a marketed drug that also opens the airways in asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Reversible asthmatic patients (>15% increase in FEV1 following 200ug salbutamol).
* FEV1 greater than or equal to 60% predicted
* Stable disease for at least the previous 3 months

Exclusion Criteria:

* Subjects requiring rescue medication on greater than 2 occasions in the 72 hours prior to screening
* Subjects with a history of pulmonary disease other than asthma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2007-05

PRIMARY OUTCOMES:
Peak and Trough (24 hour post dose) FEV1.

SECONDARY OUTCOMES:
Peak and trough (24 hour post dose) PEFR
FEV1 and PEFR measurements to 32 hours post dose.
Pharmacokinetics of PF-610,355 and salmeterol
Safety/Pharmacodynamic end points - pulse rate, blood pressure, QTcF, plasma potassium, blood glucose and AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Großhansdorf
  - Pfizer Investigational Site, Wiesbaden
- Sweden (2):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Lund
- Pfizer Investigational Site, Manchester, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7881004&StudyName=A%20Blinded%20Study%20To%20Examine%20The%20Ability%20Of%20PF-610%2C355%20To%20Open%20The%20Airways%20In%20Asthmatic%20Patients.